CLINICAL TRIAL: NCT04261790
Title: Evaluating the Effects of Ocrelizumab on B-cell Tolerance Defect in Relapsing Multiple Sclerosis
Brief Title: Effects of Ocrelizumab on B-cell Tolerance Defect in Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00230800
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ocrelizumab (Other): Patients will be treated with two courses of ocrelizumab (Ocrevus) for one year and then will stop the medication and will be monitored for the return of the disease activity. Those who experience the return of the disease activity can go back on the medication.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Patients will be treated with two courses of ocrelizumab (Ocrevus) 600mg/course, for one year and then will stop the medication and will be monitored for the return of the disease activity. Those who experience the return of the disease activity can go back on the medication.
  Other Names: Ocrevus

SUMMARY:
B-cells have an important role in the pathogenesis of multiple sclerosis (MS). Ocrelizumab, a medication that targets B-cells have been found to be highly effective in stopping the disease activity in relapsing-remitting MS.

The efficacy of ocrelizumab might be related to the specific pattern of B-cell tolerance defect in patients with MS and the potential of its normalization with treatment with ocrelizumab. By analyzing the reactivity of recombinant antibodies expressed from single B-cells, the investigators' collaborators have demonstrated that the pattern of B-cell tolerance defect is different in people with MS who only display an impaired removal of developing autoreactive B-cells in the periphery while central B-cell tolerance in the bone marrow is functional in most patients. In contrast, patients with rheumatoid arthritis (RA), type-1 diabetes (T1D) or Sjögren's syndrome (SS) show defective central and peripheral B-cell tolerance checkpoints. As a consequence, while anti-B-cell therapy does not correct defective early B-cell tolerance checkpoints in T1D and only temporarily slows down autoimmune processes before newly generated autoreactive B-cells likely induce patient relapse, the investigators postulate that the efficacy of ocrelizumab in MS may be linked to normal central B-cell tolerance and the production of a normal B-cell and T-cell compartment after ocrelizumab therapy.

In an open-label study, 10 patients with relapsing MS will be treated with two courses of ocrelizumab and will be followed clinically and radiologically for at least two and a half years. Assessment of T and B-cell phenotypes and function at baseline and 18-24 months post-B-cell depletion will be the primary outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting multiple sclerosis (RRMS) based on revised McDonald criteria
* At least one Gd-enhancing lesions on the brain or spinal cord MRI done in the prior three months OR at least one new T2/FLAIR lesion on the brain or spinal cord MRI done in the prior three months (compared to a prior MRI performed within 18 months of the most recent MRI)
* Naïve to Disease modifying therapy (DMT) or at least off these DMTs (natalizumab, fingolimod, DMF) for three months or on an injectable DMT (interferons or glatiramer acetate)
* Expanded Disability Status Scale (EDSS) score at the time of screening =<3
* Negative urine or serum pregnancy test must be available for premenopausal women and for women <12 months after the onset of menopause unless these women have undergone surgical sterilization
* Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use one method of contraception with a failure rate of <1% per year or a barrier method supplemented with spermicide. Contraception must continue for the duration of study treatment and for at least 24 weeks after the last dose of study treatment

Exclusion Criteria:

* Contraindication to treatment with an anti- cluster of differentiation antigen 20 (CD20) antibodies, including being seropositive for HBsAg
* Active hepatitis B virus infection
* Ever received B-cell depleting antibodies (rituximab, ocrelizumab, ofatumumab), alemtuzumab, daclizumab, mitoxantrone or hematopoietic stem-cell transplant
* Pregnant or lactating women
* Hypersensitivity to ocrelizumab
* Treatment with steroids in the past 30 days

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bardia Nourbakhsh, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salazar-Camelo A, Vega L, Fadlallah Y, Bou Rjeily N, Balshi A, Morris B, Ghajarzadeh M, Mowry EM, Waubant E, Nourbakhsh B. Finite-course ocrelizumab in relapsing multiple sclerosis: Results of two prospective open-label trials with matched controls. Mult Scler. 2025 Oct;31(11):1338-1347. doi: 10.1177/13524585251375350. Epub 2025 Sep 19. PMID 40970353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ocrelizumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Disease Duration [Mean (Standard Deviation); unit: years] | 2.8 (7.0)
Baseline Expanded Disability Status Scale (EDSS) [Median (Inter-Quartile Range); unit: units on a scale] — scores range from 0 to 10; the higher the score, the worse the MS-related disability
  units on a scale | 1.0 [1.0 to 1.5]
Disease-modifying Therapy (DMT) at Screening [Count of Participants; unit: Participants]
  No DMT | 8
  Glatiramer acetate | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Peripheral B-cell Tolerance Checkpoints in People With MS Before and After Ocrelizumab Therapy.
Description: By assessing the antibodies produced by isolated B-cells, changes in the frequencies (percentage) of polyreactive, and anti-nuclear clones of new emigrant/transitional and mature naive B-cells will be determined.
Time Frame: Baseline and 18-24 months
Population: Data were not collected. None of the antibodies from the immune cells were able to cloned for analysis and no data were collected from the lab samples.
Groups:
- Ocrelizumab: Ocrelizumab group
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 0

2. Primary Outcome: Change in B-cell Subpopulations
Description: Change in the frequency (percentage) of different B-cell subpopulation (assessed by flow cytometry) before and after treatment with ocrelizumab.
Time Frame: Baseline and 18-24 months
Population: as for outcome 1
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Frequency of T-cell Phenotypes
Description: Change in the frequency (percentage) of different T-cells subpopulation (assessed by flow cytometry) before and after treatment with ocrelizumab.
Time Frame: Baseline and 18-24 months
Population: as for outcome 1
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 0

4. Primary Outcome: Change in the Production of Pro Inflammatory Cytokines Produced by Activated T-cells
Description: Pro inflammatory cytokines, produced by Tregs and other T cell subsets after activating peripheral blood mononucleated cell with phorbol-12-myristate-13-acetate (PMA) and ionomycin will be measured by enzyme-linked immunosorbent assay.
Time Frame: Baseline and 18-24 months
Population: as for outcome 1
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 0

5. Primary Outcome: Change in the Production of Anti-inflammatory Cytokines Produced by Activated T-cells
Description: Anti-inflammatory cytokines, produced by Tregs and other T cell subsets after activating peripheral blood mononucleated cell with phorbol-12-myristate-13-acetate (PMA) and ionomycin will be measured by enzyme-linked immunosorbent assay
Time Frame: Baseline and 18-24 months
Population: as for outcome 1
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Patients With Return of Disease Activity
Description: Patients with the return of disease activity after the third month post-first-infusion, objectively demonstrated by development of new T2 hyperintense lesions or Gd-enhancing lesions on the MRI or a clinical relapse that is confirmed with an objective change in the neurological examination.
Time Frame: Up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 10
Participants
  Participants who did not experience the return of disease activity during the 30-month trial | 10
  Participants who experienced the return of disease activity during the 30-month trial | 0

7. Secondary Outcome: Change in Disability as Assessed by Expanded Disability Status Scale (EDSS)
Description: EDSS scores range from 0 to 10, with 0.5 steps. The higher the score, the worse the MS-related disability.
Time Frame: Screening visit and month 30 visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 10
units on a scale | -0.5 (6.0)

8. Secondary Outcome: Change in Quality of Life as Assessed by Neuro-QoL Fatigue T-score
Description: T-score (standardized scores with a mean of 50 and a standard deviation (SD) of 10). A higher Neuro-QoL T-score represents more of the concept being measured. There is no specific upper or lower limit for this scoring
Time Frame: Screening visit and month 30 visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 10
units on a scale | 2.6 (5.0)

ADVERSE EVENTS:
Time Frame: Participants received two courses of treatment with ocrelizumab six months apart. Adverse event data were collected up to 24 months after the second (last) ocrelizumab infusion.
Arm/Group | Ocrelizumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=10)
Headache (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest discomfort (Cardiac disorders) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The primary outcome measure was based on lab results; however, none of the antibodies from the immune cells were able to cloned for analysis, none of the lab samples from any participants could be analyzed, and consequently, no data for the primary outcome were generated. The study was considered completed as all participant data collection was conducted per the protocol. The failure of lab analysis affected only the primary outcome, the overall completion status is complete.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT04261790/Prot_SAP_000.pdf